CLINICAL TRIAL: NCT01193985
Title: Safety and Performance Study of TIGR Matrix Surgical Mesh in Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novus Scientific (Industry)
Responsible Party: Henrik Magnusson, Novus Scientific
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-WK-6
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: TIGR Matrix Surgical Mesh

INTERVENTIONS:
Device: TIGR Matrix Surgical Mesh — Lichtenstein repair of inguinal hernia using TIGR Matrix Surgical Mesh

SUMMARY:
This an open, uncontrolled multicenter clinical study to assess the safety and performance of the WK-6 surgical mesh in adult patients with unilateral inguinal hernia.

The primary objective is to determine the safety of the WK-6 surgical mesh. Data will be compared retrospectively with published studies on inguinal hernia mesh.

The secondary objectives are to explore the performance of the surgical mesh by measuring the pain pre and post surgery as well as a number of relevant variables for establishing the performance of the mesh. Data will be compared retrospectively with previous studies on inguinal hernia mesh with a follow-up of at least one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent
* Male, 18 years and older.
* Patients with primary unilateral inguinal hernia
* Planned surgery procedure according to Lichtenstein technique

Exclusion Criteria:

* Patients who are unwilling and/or unable to give informed consent
* Hernia strangulated or irreducible
* Recurrent Hernia
* Previous mesh surgery on the same side
* Class >IIa patients
* Unable to walk 500 meters
* BMI >30 kg/m2
* Warfarin treatment, ongoing or within two weeks of surgery.
* Peripheral artery disease
* Chronic back pain, as judged by the investigator.
* Hip joint arthrosis
* Hypermobility syndrome, as judged by the investigator.
* Constipation
* Drug or alcohol abuse
* COPD (chronic obstructive pulmonary disease)
* Patients at increased risk of death from a pre-existing concurrent illness
* Patients participating in another clinical study
* Patients who have used any other investigational drug or device within 1 month
* Patients who cannot communicate reliably with the investigator
* Patients who are unlikely to cooperate with the requirements of the study
* Patients who are employees at the investigational site; relatives or spouse of the PI.
* Patients not suitable based upon investigator decision

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events or Serious Adverse Events | 12 months
  Safety is assessed by monitoring the incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) related and unrelated to the mesh and rehabilitation. AEs and SAEs will be collected during surgery and throughout the follow up period. Possible adverse reactions with the use of any prosthesis may include but are not limited to infection, inflammation, extrusion, dhesion, fistula formation, seroma formation, hematoma, and recurrence of the hernia or tissue defect.

SECONDARY OUTCOMES:
Pain | 12 months
  The experienced pain will be measured by an ungraded Visual Analogue Scale (VAS). VAS will be assessed before the surgery and during the follow up period and elucidate the pain experienced during different conditions. A symptoms questionnaire and an analgesics diary will be used to assess the performance of the WK-6 surgical mesh for use in inguinal hernia repair.

CONTACTS AND LOCATIONS:
Overall Officials: Stellan Björck, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Kungsbacka Hospital, Kungsbacka